CLINICAL TRIAL: NCT01440257
Title: A Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Effect of CCX140-B on Albuminuria in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of CCX140-B on Urinary Albumin Excretion in Subjects With Type 2 Diabetes and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL007_140
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Nephropathy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — CCX140-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Group A) (Placebo Comparator)
  Interventions: Drug: Placebo
- Active study medication (Group B) (Experimental): CCX140-B
  Interventions: Drug: CCX140-B

INTERVENTIONS:
Drug: Placebo — Placebo capsules once daily
  Arms: Placebo (Group A)
Drug: CCX140-B — CCX140-B capsules once daily (Group B)
  Arms: Active study medication (Group B)

SUMMARY:
The purpose of this study is to evaluate the effect of treatment with CCX140-B on urinary albumin excretion in subjects with type 2 diabetes mellitus and albuminuria, as well as to study the safety and efficacy of the medication in this patient population.

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 18-75 years inclusive, with documented previously diagnosed type 2 diabetes mellitus (per American Diabetes Association [ADA] criteria), and treated with oral antidiabetic drugs
* Albumin:creatinine ratio (ACR) of 200 to 3000 mg/g creatinine, inclusive, based on two values obtained from two first morning urine samples taken on two separate days during the screening period
* Estimated glomerular filtration rate based on serum creatinine (eGFR, determined by Modification of Diet in Renal Disease [MDRD] equation) of ≥ 25 mL/min/1.73 m(2)
* Must be on a stable dose of an angiotensin-converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB) for at least 8 weeks prior to screening
* Fasting plasma glucose less than 270 mg/dL at screening

Key Exclusion Criteria:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Previous renal transplant or known non-diabetic renal disease, except related to hypertension
* Undergone renal dialysis at any time in the past
* Received chronic (more than 7 days continuously) systemic glucocorticoid or other immunosuppressive treatment within 8 weeks of screening
* Use of bardoxolone, atrasentan or other endothelin antagonist within 8 weeks of screening
* Received chronic (more than 7 days continuously) non-steroidal anti-inflammatory drug (NSAID) treatment within 2 weeks of screening
* Cardiac failure (class III or IV), history of unstable angina, symptomatic coronary artery disease, myocardial infarction or stroke within 12 weeks of screening
* Poorly-controlled blood pressure (systolic blood pressure >155 or diastolic blood pressure >95, with blood pressure measured in the seated position after at least 5 minutes of rest)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urinary albumin excretion | 84 days
  The primary efficacy objective of this study is to evaluate the effect of CCX140-B treatment on urinary albumin excretion by measuring change from baseline in 24-hour urinary albumin excretion.
Subject incidence of adverse events | 84 days
  The primary safety objective of this study is to evaluate the safety and tolerability of CCX140-B in subjects with type 2 diabetes mellitus (T2DM) with albuminuria.

SECONDARY OUTCOMES:
Change from baseline in hemoglobin A1c | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Sullivan T, Miao Z, Dairaghi DJ, Krasinski A, Wang Y, Zhao BN, Baumgart T, Ertl LS, Pennell A, Seitz L, Powers J, Zhao R, Ungashe S, Wei Z, Boring L, Tsou CL, Charo I, Berahovich RD, Schall TJ, Jaen JC. CCR2 antagonist CCX140-B provides renal and glycemic benefits in diabetic transgenic human CCR2 knockin mice. Am J Physiol Renal Physiol. 2013 Nov 1;305(9):F1288-97. doi: 10.1152/ajprenal.00316.2013. Epub 2013 Aug 28. PMID 23986513